CLINICAL TRIAL: NCT05876481
Title: Evaluation of the Acceptability, Safety, Feasibility, and Efficacy of Psilocybin-assisted Psychotherapy (PaP) for the Treatment of Post-traumatic Stress Disorder (PTSD) in Military Veterans
Brief Title: Evaluation of Psilocybin-assisted Psychotherapy (PaP) for the Treatment of Post-traumatic Stress Disorder (PTSD) in Military Veterans
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Combat Stress (Other)
Collaborators: The Watson Trust (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS-2023-002
Record Dates: First submitted 2023-04-04; First posted 2023-05-25 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: PTSD
Keywords: PTSD; Veteran; Psilocybin-assisted Psychotherapy; Feasibility trial
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Psilocybin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Psilocybin-assisted Psychotherapy (Experimental): All participants will receive 25mg psilocybin (capsule, hard, oral administration) in two 8-hour psilocybin dosing sessions, followed by Cognitive Processing Therapy.
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — Product name: Psilocybin Pharmaceutical form: capsule, hard Dose number and units: 25 mg per day (8-hour dosing session) x 2 Route of administration: oral

SUMMARY:
Post-Traumatic Stress Disorder (PTSD) is a mental health condition that occurs as a result of a traumatic experience. Symptoms include feeling anxious, flashbacks, nightmares and difficulty sleeping. Several studies indicate that psilocybin-assisted psychotherapy (PaP) may be an effective treatment for a number of mental health conditions. This has led to PaP being designated as a "breakthrough treatment" by the FDA in the US. Despite indications that PaP may hold benefits in treating individuals with posttraumatic stress disorder (PTSD), this remains to be investigated. As such, the present study aims to examine the acceptability, feasibility, safety, and efficacy of PaP (psilocybin administered with psychotherapy) in treating PTSD in military veterans.

DETAILED DESCRIPTION:
Recent studies have shown that Psilocybin-Assisted Psychotherapy (PaP) for individuals with treatment-resistant depression can result in outcomes that exceed routine psychotherapy. Psilocybin may have a catalytic effect on the psychotherapeutic process, enhancing introspection and interoception. PaP may similarly benefit the treatment of posttraumatic stress disorder (PTSD). Research indicates high treatment drop-out rates (approximately 30%) among PTSD patients, and moderate remission rates (approximately 44%) 40 months after completing treatment. Furthermore, some veterans with PTSD have poorer treatment responses than members of the general public. This suggests that alternative treatment approaches may be required to support veterans who do not benefit from standard evidence-based approaches. This study aims to explore the acceptability, feasibility, safety and efficacy of PaP for veterans with PTSD. A total of eight military veterans will be recruited. The study involves two non-directive preparatory sessions, two dosing sessions of psilocybin, followed by 12 sessions of Cognitive Processing Therapy. It is hypothesised that PaP will result in a significant reduction in PTSD symptoms, as indicated by PTSD Checklist for Diagnostic and Statistical Manual of Mental Disorders (DSM-5; PCL-5) scores from baseline to one-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-65 years
2. Fluent in English (reading and speaking)
3. Has internet access via computer or tablet
4. Is able to commit to the study visits and treatment length
5. Can provide a contact (relative, close friend, other support person) who is able to accompany the participant to dosing visits
6. Agrees to inform researchers within 48 hours of any medical treatments or procedures
7. Can swallow pills
8. Agrees to lifestyle restrictions: not to consume alcohol within 24 hours prior to dosing, and to not consume more caffeine than usual
9. Agrees to not participate in any other clinical trials for the duration of the study
10. PCL-5 score ≥33
11. At least one unsuccessful evidence-based psychotherapy/pharmacotherapy for PTSD

Exclusion Criteria:

General exclusion criteria:

1. History of poor cooperation or unreliability
2. Engaged in compensation litigation whereby financial game would be achieved from prolonged symptoms of PTSD or any other psychiatric disorders
3. Any other current problems that may interfere with participation (e.g., availability, private space for sessions at home)
4. Has hearing impairment that could interfere with ability to participate in the study
5. Is unable to provide written informed consent
6. Has known hypersensitivity or previous allergic reaction to any constituent of psilocybin
7. Pregnant or breastfeeding
8. BMI <18 or >35 or non-consent for metric to be measured during assessment visit
9. Has been diagnosed with, or has first degree relative with schizophrenia, psychotic disorder (unless substance induced or due to medical condition), or bipolar I disorder
10. Current alcohol or substance use disorder (other than caffeine or nicotine) requiring detox, or currently in withdrawal from such disorder. Exception for milder disorder if realistic plan (agreed by researcher, therapy team, and medical monitor) for successfully mitigating alcohol/substance use to prevent use from impacting participation, safety, and/or efficacy of the treatment.

    Mental health exclusion:
11. Schizophrenia spectrum or other psychotic disorders or first degree relative with such disorders (incl. major depressive disorder with psychotic features, or Bipolar I or II disorders)
12. May present serious risk to others (established via clinical interview and contact with treating psychiatrist)
13. Is likely to be re-exposed to index trauma or other significant trauma, lack social support, or lack of stable living situation

    Physical health exclusion:
14. History of myocardial infarction, angina, cerebrovascular accident, aneurysm, or pulmonary vascular disease
15. Has had Transient Ischemic Attack (TIA) within past 6 months
16. Has uncontrolled hypertension (140/90 mmHG or higher assessed on three separate occasions). Adequately controlled hypertension does not exclude participant
17. Has Wolff-Parkinson-White syndrome or other accessory pathway conditions that have not been successfully eliminated by ablation
18. History of arrhythmia, other than premature atrial contractions (PACs) or occasional premature ventricular contractions (PVCs) in the absence of ischemic heart disease, within past 12 month
19. History of risk factors for Torsade de pointes (e.g., heart failure, hypokalemia, Long QT Syndrome family history)
20. Requires use of concomitant medications that may prolong the QT/QTc interval during psilocybin dosing sessions
21. Marked Baseline prolongation of QT/corrected QT interval (QTc; e.g., repeated demonstration of a QTc interval >450ms and >460ms in females corrected by Bazett's formula). For transgender or non-binary subjects, QTc interval will be evaluated based on sex assigned at birth, unless the subject has been on hormonal treatment for five or more years.
22. History of medical condition that could make receiving a sympathomimetic drug harmful because of increased blood pressure and heart rate
23. Haptic enzymes alkaline phosphatase (ALP), alanine transaminase (ALT), Aspartate aminotransferase (AST) or Gamma-glutamyl Transferase (GGT) > three times upper limit of normal (ULN), or total bilirubin levels >2x ULN
24. Previous indication of liver or kidney damage
25. Current Hepatitis C virus (HCV) infection - Asymptomatic HCV permitted if previously undergone evaluation and treatment as needed
26. Current uncontrolled Type 2 diabetes mellitus
27. Current uncontrolled hypothyroidism
28. Current or historic glaucoma unless participation approved by an ophthalmologist
29. History of traumatic brain injury (TBI)/cognitive impairment limiting ability to engage in treatment (e.g., memory or concentration problems, impulsivity related to brain injury)
30. Current neurological illness including, but not limited to, seizure disorders, frequent migraines (or on prophylaxis for same), multiple sclerosis, movement disorders, history of significant head trauma, or central nervous system (CNS) tumour)
31. The presence of other severe acute or chronic medical condition, psychiatric condition or laboratory abnormality that may increase the risk associated with participation or may interfere with interpretation of trial results. Please note: mild, stable chronic medical problems (e.g., Type 1 or 2 Diabetes Mellitus, HIV infection, glaucoma, hypothyroidism, hepatitis C, hepatic or renal disease, etc.) may be enrolled if Investigator and research psychiatrist agree that condition(s) would not: significantly increase risk of psilocybin administration, or be likely to produce significant symptoms during the study that could interfere with participation, or be confused with side effects of Investigational Product
32. Previous use of psilocybin or other psychedelic substance (except cannabis) on more than 5 occasions and/or use of the same within the past 5 years
33. Previous use of psilocybin, methylenedioxymethamphetamine (MDMA), ketamine (or substances reportedly containing psilocybin, MDMA, or ketamine) with therapeutic aim for current PTSD diagnosis
34. Has received Electroconvulsive Therapy (ECT) within 12 weeks of enrolment
35. Requires ongoing concomitant therapy with a psychiatric medication (unless deemed acceptable by the research psychiatrist)
36. Exposure to other investigational drug/device within 30 days of enrolment

    Medication exclusion criteria:
37. Over-the-counter products intended to affect mood/anxiety
38. Efavirenz
39. Lithium
40. "Rest-Category" Antidepressants (e.g., mirtazapine, trazodone, bupropion); Exception if ≤7.5mg mirtazapine, or ≤50mg trazodone as sleeping medication
41. Antipsychotics/Neuroleptics; Exception if ≤50mg quetiapine as sleeping medication
42. Stimulants
43. The following medications are permitted if the dose is hypnotic: selective serotonin reuptake inhibitor (SSRIs); Tricyclic antidepressants (TCAs); monoamine oxidase inhibitor (MAOIs)
44. The following medications are permitted if their use is unaltered during the study: Benzodiazepines "Z-drugs" (e.g., zolpidem); Anticonvulsants; Antihistamines
45. Medications which are permitted as determined case-by-case by research psychiatrist: non-psychiatric, but mind-altering medication (e.g., morphine, dexamethasone, etc.).
46. Not to be used 72hrs prior to psilocybin dosing session: Sildenafil (Viagra), tadalafil, or similar medications
47. Not to be used on dosing days and research psychiatrist discretion: Medical cannabis

    Risk exclusion criteria:
48. Current suicidal ideation/intent/action
49. Previous (within previous 6 months) suicidal ideation/intent/action
50. Current and previous deliberate self-harm

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Symptoms of PTSD measured using the Posttraumatic Stress Disorder Checklist For DSM-5 (PCL- PTSD symptoms | Change from baseline PCL-5 score at one month follow up
  Symptoms of PTSD measured using the Posttraumatic Stress Disorder Checklist For DSM-5 (PCL- 5). Scores range from 0-80, with a higher score indicated a worse outcome.

SECONDARY OUTCOMES:
Core features of PTSD and complex PTSD measured using the International Trauma Questionnaire (ITQ) | Change from baseline ITQ score at one month follow up
  Scores range from 0 to 48 with a higher score indicating a worse outcome.
Difficulties with anger measured using the Dimensions of Anger Reactions (DAR-5) | Change from baseline DAR-5 score at one month follow up
  Scores range from 5-25, with a higher score indicating a worse outcome.
Depression symptoms measured using the Patient Health Questionnaire (PHQ-9) | Change from baseline PHQ-9 score at one month follow up
  Scores range from 0-27, with a higher score indicating a worse outcome.
General anxiety symptoms measured using the Generalised Anxiety Disorder (GAD-7) | Change from baseline GAD-7 score at one month follow up
  Scores range from 0-14, with a higher score indicating a worse outcome.
Mental wellbeing measured using the Short Warwick-Edinburgh Mental Wellbeing Scale (SWEMWBS) | Change from baseline SWEMWBS score at one month follow up
  Scores range from 7-35, with a lower score indicating a worse outcome.
Perceived social support measured using the Oslo Social Support Scale | Change from baseline OSS score at one month follow up
  Scores range from 3-14, with a higher score indicating a worse outcome.
Challenging aspects of experiences with psilocybin measured using the Challenging Experience Questionnaire | Administered at the end of dosing session one, week 4
  Scores range from 5-25, with a higher score indicating a worse outcome.
Challenging aspects of experiences with psilocybin measured using the Challenging Experience Questionnaire | Administered at the end of dosing session two, week 5
  Measures a phenomenological profile of experiences with scores not indicative of more or less strongly challenging experiences.

OTHER OUTCOMES:
Semi-structured qualitative interviews | Consenting participants will be contacted at one-month follow up.
  Intervention acceptability and experiences of the study will be measured using semi-structured qualitative interviews
Adverse Experiences in Psychotherapy | Treatment end (at CPT session 12), week 8
  Experiences that may occur in therapy measured using the Adverse Experiences in Psychotherapy to assess feasibility
Retention rate | Study end (approximately 2 years)
  Feasibility endpoint
Did Not Attend (DNA) rate | Study end (approximately 2 years)
  Feasibility endpoint
Recruitment of target sample size (n = 8) | Study end (approximately 2 years)
  Feasibility endpoint
Incidence of adverse events across the duration of the study | Study end (approximately 2 years)
  Safety endpoint, calculated as total number of adverse events reported across the study. Adverse events as defined in the study protocol.
Hazardous and harmful alcohol use measured using the Alcohol Use Disorder Identification Test | Baseline
  Background measure. Scores range from 0-40, with a higher score indicating a worse outcome.
Possible drug-related problems measured using the Drug Use Disorders Identification Test | Baseline
  Background measure. Scores range from 0-44, with a higher score indicating a worse outcome.
Difficulties with moral injury in relation to a potentially morally injurious event measured using the Moral Injury Outcome Scale (MIOS) | Baseline
  Background measure. Scores range from 0-56, with a higher score indicating a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dominic Murphy, Principal Investigator — Combat Stress
Locations (1):
- Combat Stress, Leatherhead, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carhart-Harris R, Giribaldi B, Watts R, Baker-Jones M, Murphy-Beiner A, Murphy R, Martell J, Blemings A, Erritzoe D, Nutt DJ. Trial of Psilocybin versus Escitalopram for Depression. N Engl J Med. 2021 Apr 15;384(15):1402-1411. doi: 10.1056/NEJMoa2032994. PMID 33852780
- [Background] Davis AK, Barrett FS, May DG, Cosimano MP, Sepeda ND, Johnson MW, Finan PH, Griffiths RR. Effects of Psilocybin-Assisted Therapy on Major Depressive Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2021 May 1;78(5):481-489. doi: 10.1001/jamapsychiatry.2020.3285. PMID 33146667
- [Background] Dos Santos RG, Hallak JEC. Therapeutic use of serotoninergic hallucinogens: A review of the evidence and of the biological and psychological mechanisms. Neurosci Biobehav Rev. 2020 Jan;108:423-434. doi: 10.1016/j.neubiorev.2019.12.001. Epub 2019 Dec 3. PMID 31809772
- [Background] Nichols DE. Psychedelics. Pharmacol Rev. 2016 Apr;68(2):264-355. doi: 10.1124/pr.115.011478. PMID 26841800
- [Background] Cloitre M, Stolbach BC, Herman JL, van der Kolk B, Pynoos R, Wang J, Petkova E. A developmental approach to complex PTSD: childhood and adult cumulative trauma as predictors of symptom complexity. J Trauma Stress. 2009 Oct;22(5):399-408. doi: 10.1002/jts.20444. Epub 2009 Sep 30. PMID 19795402
- [Background] Morina N, Wicherts JM, Lobbrecht J, Priebe S. Remission from post-traumatic stress disorder in adults: a systematic review and meta-analysis of long term outcome studies. Clin Psychol Rev. 2014 Apr;34(3):249-55. doi: 10.1016/j.cpr.2014.03.002. Epub 2014 Mar 14. PMID 24681171
- [Background] Kitchiner NJ, Roberts NP, Wilcox D, Bisson JI. Systematic review and meta-analyses of psychosocial interventions for veterans of the military. Eur J Psychotraumatol. 2012;3. doi: 10.3402/ejpt.v3i0.19267. Epub 2012 Dec 5. PMID 23233869
- [Background] Straud CL, Siev J, Messer S, Zalta AK. Examining military population and trauma type as moderators of treatment outcome for first-line psychotherapies for PTSD: A meta-analysis. J Anxiety Disord. 2019 Oct;67:102133. doi: 10.1016/j.janxdis.2019.102133. Epub 2019 Aug 18. PMID 31472332